CLINICAL TRIAL: NCT01040234
Title: Ultrasound-guided Bilateral Dual Transversus Abdominis Plane (BD-TAP) Block: Description of a Novel Four-point Ultrasound-guided TAP Block Approach
Brief Title: Bilateral Dual TAP Block: Description of a Novel Four-point Approach
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Kenneth Jensen, MD, BBA, MD, BBA, Bispebjerg Hospital
Other Study IDs: BBH_Z-Regional-001
Record Dates: First submitted 2009-12-17; First posted 2009-12-29 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; abdominal surgery; bilateral dual TAP block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Active pain treatment: Bilateral dual TAP block
  Interventions: Procedure: Bilateral dual TAP block

INTERVENTIONS:
Procedure: Bilateral dual TAP block — Bupivacaine 2.5 mg/ml 15 ml per injection. 4 injections per patient according to dual TAP block procedure
  Other Names: Marcain; TAP block

SUMMARY:
A prospective study of 30 patients with severe postoperative pain following abdominal surgery, in which the dual TAP block technique has been used successfully to achieve pain relief. A description of ultrasound technique, effectiveness, duration and potential side effects of the pain treatment, with possible recommendations for future use.

DETAILED DESCRIPTION:
This prospective cohort study is designed to describe a novel ultrasound-guided bilateral dual transversus abdominis plane (BD-TAP) block and to evaluate the postoperative analgesic efficacy in a selection of patients having undergone major abdominal surgery under general anaesthesia where neuraxial anaesthesia and/or intravenous administration of analgesics had failed or was unwanted by the patient, or if the placement of an epidural catheter was deemed impossible by the anaesthetist in charge. 30 consecutive patients planned for the study. BD-TAP to be performed bilaterally with a high frequency linear ultrasound probe, with bupivacaine. Success rate, decline in VAS score, postoperative demand of opioids and block performance time to be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain VAS >5 following abdominal surgery, in which conventional pain treatment or epidural block is either ineffective or contraindicated

Exclusion Criteria:

* Hypersensitivity to local anaesthetics

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with postoperative pain following abdominal surgery that do not respond to moderate doses of opioid analgesics or patients with failed epidurals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pain VAS after the intervention compared to pre-intervention VAS | 10-20 minutes after intervention

SECONDARY OUTCOMES:
Pain medication required following intervention | First 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jens N Børglum, MD, PhD, Principal Investigator — Dept Z, Bispebjerg Hospital
Locations (1):
- Dept Z, Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark